CLINICAL TRIAL: NCT00743392
Title: HPV Infections in Older Women
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Rachel Winer, Assistant Professor, University of Washington
Other Study IDs: 34339-A
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal swab samples for HPV DNA testing
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine risk factors for HPV infections in 25 to 65 year old women who report having used internet dating websites in the past year.

DETAILED DESCRIPTION:
Whether older women are susceptible to acquiring new, persistent high-risk (HR) HPV infections from new sex partners is largely unknown. This is a longitudinal study of predictors of HR HPV infections in two populations of women aged 25 to 44 and 45 to 65 who have used internet dating websites in the past year. 300 women will be recruited and mailed kits for self-collecting vaginal specimens for HPV DNA testing. Women will self-collect four sets of vaginal specimens four months apart, and complete sexual behavior questionnaires at the time of each self-collection. We will identify behavioral and health predictors of type-specific HR HPV infections, predictors of repeatedly-detected HR HPV infections, and evaluate study participants' experiences with self-collecting vaginal specimens and attitudes towards HPV vaccination and cervical cancer screening. This information is important for developing guidelines for HPV vaccine implementation and cervical cancer screening guidelines in populations of older women.

ELIGIBILITY:
Inclusion Criteria:

* Have had sex with men
* Have used the internet to search for romantic partners in the past year (e.g. posted or responded to an ad on an internet dating website or social networking website)

Exclusion Criteria:

* Pregnant, breastfeeding, or planning a pregnancy in the next 6 months
* Hysterectomy

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 to 65 year old women who date online
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
High-risk HPV DNA | Every 4 months for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Winer, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- See also: HPV study website — http://depts.washington.edu/hpvstudy